CLINICAL TRIAL: NCT04526704
Title: A Phase 4, Multicenter Study to Evaluate Discontinuation and Re-Treatment in Subjects With Tenosynovial Giant Cell Tumor (TGCT) Previously Treated With Pexidartinib
Brief Title: Study to Evaluate Discontinuation and Re-Treatment in Participants With Tenosynovial Giant Cell Tumor (TGCT) Previously Treated With Pexidartinib
Acronym: PLX3397
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL3397-A-U4003; 2020-000192-20 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Tenosynovial Giant Cell Tumor
Keywords: Tenosynovial Giant Cell Tumor; Pexidartinib; TURALIO™️; PLX3397
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Continuation Cohort (Experimental): Previously-treated participants with TGCT continuing their current dose of pexidartinib treatment.
  Interventions: Drug: Pexidartinib
- Treatment-Free/Re-Treatment Cohort (Experimental): Previously-treated participants with TGCT who discontinue pexidartinib treatment (Treatment-Free Period) and had the option to resume pexidartinib treatment at dose at completion of prior study (Re-Treatment Period).
  Interventions: Drug: Pexidartinib

INTERVENTIONS:
Drug: Pexidartinib — 200 mg capsules administered orally twice daily on an empty stomach (at least 1 hour before or at least 2 hours after a meal or snack)
  Other Names: TURALIO™️; PLX3397

SUMMARY:
This study is designed to evaluate the discontinuation/re-treatment of pexidartinib therapy in previously treated participants with tenosynovial giant cell tumor (TGCT).

DETAILED DESCRIPTION:
This multicenter study in previously pexidartinib-treated participants with TGCT will provide the Investigators and participants the option at Screening to either continue pexidartinib treatment (Treatment Continuation Cohort) or discontinue treatment with the possibility of re-initiating pexidartinib treatment (Treatment-Free/Re-Treatment Cohort).

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and on pexidartinib treatment in one of the following studies: Study PLX108-10 (ENLIVEN), Study PLX108-01, Study PL3397-A-A103 or Study PL3397-A-U126.
* Willing and able to complete the PROMIS Physical Function Scale and EQ-5D-5L throughout the study.
* Willing and able to provide written informed consent prior to any study-related procedures and to comply with all study requirements.
* Females of reproductive potential must have a negative urine pregnancy test at Screening/Baseline (to be confirmed by a serum pregnancy test taken on the last treatment visit of their prior study). They are advised to use an effective, non-hormonal method of contraception during treatment with pexidartinib and for 1 month after the last dose. Males with female partners of reproductive potential should be advised to use an effective method of contraception during treatment with pexidartinib and for 1 month after the last dose. Female partners of male patients should concurrently use effective contraceptive methods (hormonal or non-hormonal).

Note: A female is considered of reproductive potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy) with a confirmed by follicle stimulating hormone (FSH) test level >40 mIU/mL.

* Male participants must not freeze or donate sperm starting at Screening and throughout the study period, and for at least 5 half-lives or 1 month after the final study drug administration, whichever is longer. Female participants must not donate, or retrieve for their own use, ova from the time of Screening and throughout the study treatment period, and for at least 1 month or 5 half-lives after the final study drug administration, whichever is longer.

Exclusion Criteria:

* Participant has a clinically significant abnormality identified by the Investigator at Screening on physical examination, laboratory tests, or electrocardiogram (ECG) which, in the judgement of the Investigator, would preclude the participant's safe completion of the study.
* Exposure to another investigational drug or current participation in other therapeutic investigational procedures, besides pexidartinib studies, within 1 month prior to start of study treatment. Any known contraindication to treatment with, including hypersensitivity to, the study drug(s) or excipients in pexidartinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Daiichi Sankyo
Locations (16):
- United States (7):
  - Honor Health, Scottsdale, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
- Magyar Honvedseg Egeszsegugyi Kozpont, Budapest, Hungary
- Italy (2):
  - Rizzoli-Istituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCC Istituto Nazionale dei Tumori, Milan
- Leiden University Medical Center (LUMC), Leiden, Netherlands
- Spain (2):
  - Hospital Sant Pau, Barcelona
  - Hospital Virgen del Rocio, Seville
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study.
Pre-assignment Details: As specified in the protocol, the study analysis was conducted based on 2 cohorts: Treatment Continuation Cohort and Treatment-Free/Re-Treatment Cohort.
Groups:
- Treatment Continuation Cohort: Previously-treated participants with TGCT who continued their current dose of pexidartinib treatment.
- Treatment-Free/Re-Treatment Cohort: Previously-treated participants with TGCT who discontinued pexidartinib treatment (Treatment-Free Period) and had the option to resume pexidartinib treatment at dose of completion of prior study (Re-Treatment Period).
Period: Overall Study
Arm/Group | Treatment Continuation Cohort | Treatment-Free/Re-Treatment Cohort
Started | 21 | 11
Resumed Pexidartinib Treatment | 0 | 3
Completed | 17 | 11
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Continuation Cohort | Treatment-Free/Re-Treatment Cohort | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (15.7) | 51.9 (15.2) | 48.2 (15.5)
Age, Customized [Count of Participants; unit: Participants]
  18 to 40 years | 7 | 1 | 8
  41 to 64 years | 12 | 8 | 20
  65 to 74 years | 1 | 1 | 2
  75 to 84 years | 1 | 1 | 2
  ≥ 85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  White | 19 | 8 | 27
  Not collected per local regulations | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Free Participants at 12 Months In The Treatment-free/Re-treatment Cohort
Description: Participants who were not remaining treatment-free were defined as either participants who resumed pexidartinib treatment, death (any cause) or who were receiving systemic therapy or undergoing surgery for the treatment of TGCT, whichever occurs first. The number of participants who remained treatment-free at Month 12 is reported.
Time Frame: Baseline up to 12 months after last participant enrolled in Cohort
Population: The number of treatment-free participants was assessed in participants with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 11
Participants | 8

2. Primary Outcome: Number of Treatment-Free Participants at 24 Months In The Treatment-free/Re-treatment Cohort
Description: Participants who were not remaining treatment-free were defined as either participants who resumed pexidartinib treatment, death (any cause) or who were receiving systemic therapy or undergoing surgery for the treatment of TGCT, whichever occurs first. The number of participants who remained treatment-free at Month 24 is reported.
Time Frame: Baseline up to 24 months after last participant enrolled in Cohort
Population: The number of treatment-free participants was assessed in participants with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 11
Participants | 8

3. Secondary Outcome: Change From Baseline in PROMIS Physical Function Total Overall Score In The Treatment Continuation and Treatment-free/Re-Treatment Cohorts
Description: The PROMIS Physical Function Total Overall Score (includes 11 upper extremity questions and 13 lower extremity questions) ranges from 24 to 120, with each individual question being rated on a 5-point rating scale (where 1 is unable to do and 5 is without any difficulty). Higher PROMIS Physical Function Total Overall Scores indicate a better health state. The change from baseline in PROMIS Physical Function Total Overall Scores is being reported.
Time Frame: Baseline up to Month 24
Population: PROMIS Physical Function was assessed in participants with available data in the Evaluable Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Continuation Cohort | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 16 | 7
score on a scale | -2.78 (6.42) | -1.93 (4.80)

4. Secondary Outcome: Change From Baseline in EQ-5D-5L Scale Score In The Treatment Continuation and Treatment-free/Re-Treatment Cohorts
Description: The EQ-5D-5L questionnaire assessed a participant's mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The overall health is rated on a scale from 0 to 100, where 0 is worst health you can imagine and 100 is best health you can imagine. The change from baseline in EQ-5D-5L Scale Score is being reported.
Time Frame: Baseline up to Month 24
Population: EQ-5D-5L was assessed in participants with available data in the Evaluable Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Continuation Cohort | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 16 | 7
score on a scale | -2.4 (13.53) | 3.4 (7.59)

5. Secondary Outcome: Number of Participants With and Without Progressive Disease
Description: Tumors were assessed based on the RECIST criteria. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; ≥30% increase in volume relative to lowest score during the study whether at baseline or some other visit.
Time Frame: Month 18 (Re-treatment Period of the Treatment-free/Re-treatment Cohort), Month 24 (Treatment Continuation Cohort)
Population: Tumor assessments were analyzed in participants with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continuation Cohort | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 16 | 3
Participants
  Not progressive | 16 | 0
  Progressive disease | 0 | 1
  Not evaluable | 0 | 0

6. Secondary Outcome: Number of Participants Who Reported Treatment-Emergent Adverse Events (TEAEs) In The Treatment Continuation Cohort
Description: Treatment-emergent adverse events (TEAEs) were defined as new adverse events (AEs) or pre-existing conditions that worsen in CTCAE grade after the first dose of study drug and up to 30 days after last dose of study drug.
Time Frame: Baseline up to 30 days after the start of re-treatment or end of study (whichever occurs first), up to 24 months
Population: Treatment-emergent adverse events were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continuation Cohort
Number analyzed (Participants) | 21
Participants | 19

7. Secondary Outcome: Number of Participants Who Reported Treatment-Emergent Adverse Events (TEAEs) In The Re-Treatment Period of the Treatment-free/Re-Treatment Cohort
Description: as for outcome 6
Time Frame: Baseline up to 30 days after the start of re-treatment or end of study (whichever occurs first), up to 24 months
Population: Treatment-emergent adverse events were assessed in participants with available data in the Safety Analysis Set .
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 3
Participants | 3

8. Secondary Outcome: Number of Patients Reporting AEs (Treatment-free)
Description: Adverse events (AEs) were defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product and that does not necessarily have to have a causal relationship with this treatment. Participants who were not remaining treatment-free were defined as either participants who resumed pexidartinib treatment, death (any cause) or who were receiving systemic therapy or undergoing surgery for the treatment of TGCT, whichever occurs first.
Time Frame: Baseline up to 30 days after the start of re-treatment or end of study (whichever occurs first), up to 24 months
Population: Adverse events were assessed in the Safety Analysis Set in participants with available data in the Treatment-free Period of the Treatment-Free/Re-Treatment Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Free/Re-Treatment Cohort
Number analyzed (Participants) | 11
Participants
  Any Grade AE | 7
  Any Grade Musculoskeletal/Tissue Disorders | 6
  Any Grade Arthralgia | 2
  Any Grade Back pain | 2
  Any Grade Intervertebral disc protrusion | 1
  Any Grade Joint swelling | 1
  Any Grade Musculoskeletal pain | 1
  Any Grade Pain in extremity | 1
  Any Grade Metabolism and Nutrition Disorders | 3
  Any Grade Hypercholesterolaemia | 2
  Any Grade Hypertriglyceridaemia | 2
  Any Grade General Disorders & Site Conditions | 2
  Any Grade Asthenia | 1
  Any Grade Oedema peripheral | 1
  Any Grade Infections and Infestations | 2
  Any Grade Cellulitis | 1
  Any Grade COVID-19 | 1
  Any Grade investigations | 2
  Any Gr Blood creatinine phosphokinase increased | 2
  Any Grade Blood uric acid increased | 1
  Any Renal and Urinary Disorders | 2
  Any Renal colic | 1
  Any Grade Urinary retention | 1
  Any Grade Injury, Poisoning & Procedural Issues | 1
  Any Grade Animal bite | 1
  Any Grade Neoplasms Benign, Malignant & Other | 1
  Any Grade Lipoma | 1
  Any Grade Nervous System Disorders | 1
  Any Grade Sciatica | 1
  Any Grade Skin and Subcutaneous Tissue Disorders | 1
  Any Grade Urticaria | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from baseline up to 30 days after the start of re-treatment or end of study (whichever occurs first), up to 24 months.
Description: TEAEs observed in the Treatment Continuation Cohort and the Re-Treatment Period of the Treatment-free/Re-Treatment Cohort are reported. AEs from the Treatment-free Period of the Treatment-free/Re-Treatment Cohort were captured and are reported as well.
Groups:
- Re-Treatment Period of Treatment-Free/Re-Treatment Cohort: Previously-treated participants with TGCT who discontinued pexidartinib treatment (Treatment-Free Period) and had the option to resume pexidartinib treatment at dose of completion of prior study (Re-Treatment Period).
- Treatment-Free Period of Treatment-Free/Re-treatment Cohort: Previously-treated participants with TGCT who discontinued pexidartinib treatment (Treatment-Free Period) and reported adverse events.
Arm/Group | Treatment Continuation Cohort | Re-Treatment Period of Treatment-Free/Re-Treatment Cohort | Treatment-Free Period of Treatment-Free/Re-treatment Cohort
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/3 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/3 | 0/11
Other Adverse Events (participants affected / at risk) | 19/21 | 3/3 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Continuation Cohort (N=21) | Re-Treatment Period of Treatment-Free/Re-Treatment Cohort (N=3) | Treatment-Free Period of Treatment-Free/Re-treatment Cohort (N=11)
Creutzfeldt-Jakob disease (Infections and infestations) | 1 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Continuation Cohort (N=21) | Re-Treatment Period of Treatment-Free/Re-Treatment Cohort (N=3) | Treatment-Free Period of Treatment-Free/Re-treatment Cohort (N=11)
COVID-19 (Infections and infestations) | 7 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Blood creatinine phosphokinase increased (Investigations) | 8 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 3 | 1 | 1
Fatigue (General disorders) | 3 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Intevertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT04526704/Prot_SAP_000.pdf